CLINICAL TRIAL: NCT04882293
Title: Confirmatory Study of the Efficacy and Safety of the Fixed-dose Combination Atorvastatin / Fenofibrate Versus Atorvastatin on the Lipid Profile of Patients With Type 2 Diabetes (T2D) and Dyslipidaemia (DLP).
Brief Title: Efficacy and Safety of the Fixed-dose Combination Atorvastatin/Fenofibrate vs Atorvastatin in Patients With T2D and DLP.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SIL-30301-III-20(1)
Record Dates: First submitted 2021-04-29; First posted 2021-05-11 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Dyslipidemia Associated With Type II Diabetes Mellitus
Keywords: Dyslipidemia; Type 2 diabetes; Hypertriglyceridemia; Lipid profile
MeSH Terms: conditions — Dyslipidemias; Diabetes Mellitus, Type 2; Hypertriglyceridemia | interventions — Atorvastatin; Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Atorvastatin / Fenofibrate in fixed dose (Experimental): Group A: Atorvastatin / Fenofibrate in fixed dose Pharmaceutical Form: Tablets Dosage: 20 mg /160 mg Adminstration way: Oral
  Interventions: Drug: Atorvastatin 20 mg / Fenofibrate 160 mg in fixed dose
- Group B: Atorvastatin (Lipitor ®) (Active Comparator): Group B: Atorvastatin (Lipitor ®) Pharmaceutical Form: Tablets Dosage: 20 mg Adminstration wat: Oral
  Interventions: Drug: Atorvastatin (Lipitor ®)

INTERVENTIONS:
Drug: Atorvastatin 20 mg / Fenofibrate 160 mg in fixed dose — 1 tablet once a day, 20 mg /160 mg, Orally
  Other Names: ATV / FENO
  Arms: Group A: Atorvastatin / Fenofibrate in fixed dose
Drug: Atorvastatin (Lipitor ®) — 1 tablet once a day, 20 mg, Orally
  Other Names: ATV (Lipitor ®)
  Arms: Group B: Atorvastatin (Lipitor ®)

SUMMARY:
Phase IIIb, randomized, longitudinal, prospective, multicenter study to evaluate the efficacy and safety of the fixed-dose combination atorvastatin / fenofibrate versus atorvastatin on the lipid profile of patients with type 2 diabetes and dyslipidemia.

DETAILED DESCRIPTION:
To assess the efficacy and safety of the fixed-dose combination atorvastatin / fenofibrate versus atorvastatin on the lipid profile of patients with type 2 diabetes and dyslipidemia. Assessing the magnitude of change in lipid profile numbers. And describing the effect on anthropometric, biochemical and clinical indicators, as well as events and adverse reactions that may occur. In patients diagnosed with type 2 diabetes and dyslipidemia (triglycerides> 150 mg / dl, LDL (Low density lipoprotein) cholesterol> 100 mg / dl) and who require pharmacological treatment for lipid control.

ELIGIBILITY:
Inclusion Criteria:

* That the subject agrees to participate in the study and gives their informed consent in writing.
* Both genres.
* Age 18 to 75 years old.
* Diagnosis of type 2 diabetes mellitus with adequate glycemic control defined by HbA1c ≤ 7.5% at the time of selection.
* Diagnosis of dyslipidemia prior to the start of the study (LDL cholesterol> 100 mg / dl and triglycerides> 150 mg / dl).
* Willing to avoid sexual contact or to use a barrier method of contraception while conducting the study.

Exclusion Criteria:

* The drug is contraindicated for medical reasons.
* Consumption of oral contraceptives, cyclosporine or strong cytochrome p450 (CYP) 3A4 inhibitors, protease inhibitors, erythromycin and azoles.
* Patients with Type 1 Diabetes Mellitus.
* Acute or Severe renal dysfunction (glomerular filtration <30 ml / min / 1.72 m2).
* History of chronic liver disease or ALT and / or AST ≥ 2 times the upper limit of normal, or GGT ≥3 times the upper limit of normal.
* Chronic or acute pancreatitis except for acute pancreatitis due to severe hypertriglyceridemia (defined by the presence of triglycerides> 1000 mg / dl and / or milky plasma, in the absence of other etiological factors of pancreatitis).
* Patients with active gallbladder disease (defined as acute or chronic gallbladder disorders associated with clinical signs or symptoms).
* Patient with a history or presence of myopathies.
* Pregnant or lactating women.
* Known contraindication or hypersensitivity to the use of any of the components of the investigational drug.
* The patient is participating in another clinical study involving an investigational treatment or participated in one in the previous 4 weeks.
* At the medical discretion, a disease that affects the prognosis and prevents outpatient management, for example, but not restricted to: end-stage cancer, kidney, heart, respiratory or liver or mental failure or with scheduled surgical or hospital procedures.
* Be a patient with a working relationship with the principal investigator or the research center or prisoner.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Magnitude of change in lipid profile figures. | Baseline, 2 and 4 months.
  To assess the magnitude of change in lipid profile figures (Lp [a], LDL, and triglycerides) at 2 and 4 months with respect to their baseline measurement and between treatment groups.
Proportion of subjects achieving triglyceride levels <150 mg /dL. | 4 months
  Describe the proportion of subjects who achieved triglyceride levels <150 mg / dL at the end of treatment.
Describe the proportion of subjects who reduced levels of LDL cholesterol | Baseline and 4 months.
  Describe the proportion of subjects who reduced levels of LDL cholesterol, under 30% compare to the baseline value.

SECONDARY OUTCOMES:
Impact on anthropometric indicators (Weight) | Baseline and 4 Months
  Describe changes in weight (kg) measurements from baseline to the end of the study (4 months).
Impact on anthropometric indicators body mass index (BMI) | Baseline and 4 months
  Describe changes in BMI (kg/m2) from baseline to the end of the study (4 months)
Impact on anthropometric indicators (Waist circumference) | Baseline and 4 months
  Describe changes in waist circumference (cm) from baseline to the end of the study (4 months).
Impact on liver function with aspartate aminotransferas (AST) | Baseline and 4 months
  Describe the changes in AST (mg/dL) concentration, between baseline and the end of the study.
Impact on liver function with Alanine Aminotransferase (ALT) | Baseline and 4 months
  Describe the changes in ALT (mg/dL) concentration, between baseline and the end of the study.
Impact on Glycosylated hemoglobin (HbA1c) | Baseline and 4 months
  Describe the changes in HbA1c percentage from baseline to the end of the study (4 months).
Impact on glucose levels | Baseline and 4 months
  Describe the changes in glucose levels (mg/dL) from baseline to the end of the study (4 months).
Impact on Blood pressure | Baseline and 4 months
  Describe the changes in blood pressure (mm Hg) from baseline to the end of the study (4 months). impact on clinical indicators (Blood pressure, Heart rate, Respiratory rate).
Impact on heart rate | Baseline and 4 months
  Describe the changes in heart rate (beats per minute) from baseline to the end of the study (4 months).
Impact on respiratory rate | Baseline and 4 months
  Describe the changes in respiratory rate (Pulses per minute) from baseline to the end of the study (4 months).
Events and adverse reactions presented. | 4 months
  Proportion of events and adverse reactions presented during 4 months of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto J Zamora Muciño-Arroyo, M.D, Principal Investigator — Investigación Biomédica para el Desarrollo de Fármacos S.A. de C.V. (BIOMED-AGS); Joel Rodríguez Saldaña, M.D, Principal Investigator — Resultados médicos, desarrollo e investigación SC (REMEDI); Francisco G Padilla Padilla, M.D, Principal Investigator — Independent; Juan A Peraza Zaldivar, M.D, Principal Investigator — Investigación Biomédica para el Desarrollo de Fármacos S.A. de C.V. (BIOMED-GDL); Luis M Román Pintos, PhD, Principal Investigator — Hospital Hispano S.A de C.V
Locations (1):
- Laboratorio Silanes, S.A. de C.V., Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Escobedo-de la Pena J, de Jesus-Perez R, Schargrodsky H, Champagne B. [Prevalence of dyslipidemias in Mexico city and Its relation to other cardiovascular risk factors. Results from the CARMELA study]. Gac Med Mex. 2014 Mar-Apr;150(2):128-36. Spanish. PMID 24603993
- [Background] Harivenkatesh N, David DC, Haribalaji N, Sudhakar MK. Efficacy and safety of alternate day therapy with atorvastatin and fenofibrate combination in mixed dyslipidemia: a randomized controlled trial. J Cardiovasc Pharmacol Ther. 2014 May;19(3):296-303. doi: 10.1177/1074248413518968. Epub 2014 Feb 10. PMID 24516261
- [Background] Lella M, Indira K. A comparative study of efficacy of atorvastatin alone and its combination with fenofibrate on lipid profile in type 2 diabetes mellitus patients with hyperlipidemia. J Adv Pharm Technol Res. 2013 Jul;4(3):166-70. doi: 10.4103/2231-4040.116778. PMID 24083205
- [Background] Athyros VG, Papageorgiou AA, Athyrou VV, Demitriadis DS, Kontopoulos AG. Atorvastatin and micronized fenofibrate alone and in combination in type 2 diabetes with combined hyperlipidemia. Diabetes Care. 2002 Jul;25(7):1198-202. doi: 10.2337/diacare.25.7.1198. PMID 12087019
- [Derived] Padilla-Padilla FG, Ruiz-Bernes LN, Roman-Pintos LM, Peraza-Zaldivar JA, Sander-Padilla JG, Lugo-Sanchez LA, Rios-Brito KF, Arguedas-Nunez MM, Flores-Huanosta D, Gonzalez-Canudas J. Efficacy and Safety of the Fixed-Dose Combination of Atorvastatin/Fenofibrate Versus Atorvastatin on the Lipid Profile of Patients with Type 2 Diabetes and Dyslipidemia. Cardiol Ther. 2025 Jun;14(2):297-314. doi: 10.1007/s40119-025-00410-y. Epub 2025 May 5. PMID 40323331
- See also: NOM. 037-SSA2-2012 para la prevención, tratamiento y control de las dislipidemias. México: Diario Oficial de la Federación. 2012;13. — https://www.dof.gob.mx/nota_detalle.php?codigo=5259329&fecha=13/07/2012